CLINICAL TRIAL: NCT02250040
Title: Development and Assessment of a New Physiotherapy Protocol for Gait Recovery After Stroke Based on Clinical and Functional Criteria
Brief Title: Effect of a Physiotherapy Protocol for Gait and Functional Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, M Luz Sanchez, DPT, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/0417
Record Dates: First submitted 2014-04-02; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Physiotherapy; Functional Recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Conventional physiotherapy for stroke.
  Interventions: Other: Conventional physiotherapy
- Target group (Experimental): Techniques based on patients' functional level were added.
  Interventions: Other: Conventional physiotherapy; Other: Techniques based on patients' functional level were added.

INTERVENTIONS:
Other: Conventional physiotherapy — Physiotherapy techniques that included muscle training, stretching and endurance.
Other: Techniques based on patients' functional level were added. — The added techniques aimed to improve balance and movement dissociation.
  Arms: Target group

SUMMARY:
The purpose of this study was to identify and evaluate the effect of a new protocol of physiotherapy to retrain walking ability after stroke in subjects older than fifty-five. This protocol was composed of specific, clearly defined and reproducible techniques, based on clinical and functional criteria.

DETAILED DESCRIPTION:
Stroke is a major cause of morbidity and mortality in adults and the leading cause of disability in all developed countries. Its incidence is approximately one million per year in the European Union.

It produces a huge social impact, not only because of mortality but also by the high demand for health and social services that involve its disabling effects on more than thirty thousand Spanish every year. Hemiplegia is the most common physical consequence of stroke and it is defined as the complete paralysis of the upper and lower extremities of one body side. However, other consequences as perceptual, cognitive, sensory and communication problems should be considered in the physiotherapy treatment.

Age is the most important risk indicator of stroke as it represents an exponential increase in incidence. After the age of 55 the risk doubles for every decade and triples at 80. After rehabilitation, most people who have suffered a stroke get to walk independently or with some technical help, but approximately 50-60% continue to have a certain degree of motor impairment and approximately 50% are, at least in part, dependent for daily life activities. Therefore, gait recovery is one of the main objectives in the rehabilitation process of stroke survivors.

Regarding the process of rehabilitation after stroke, currently, there is insufficient evidence to conclude that any of the physical therapy approaches is more effective to promote recovery of lower limb function or postural control than any other. Thus, future research should focus on determining the effectiveness of individual techniques clearly described and specific treatments for each problem regardless of their approach. Furthermore, after reviewing the different approaches of physiotherapy rehabilitation after stroke, no physiotherapy treatment protocols based on clinical status of the patient have been found. Instead, vague and general instructions are given, so it is necessary to clarify what to do, when and what is the effectiveness of these techniques.

On the other hand, studies have scarcely taken into account the special characteristics of the elderly as a population group so involved in this pathology.

This study aims at addressing these issues, since its main objective is to identify and evaluate the effect of a protocol of physiotherapy to retrain walking ability after stroke in patients older than fifty-five, composed of specific, clearly defined and reproducible techniques, based on clinical and functional criteria.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered a single stroke episode with residual hemiparesis
* Being candidate to begin a rehabilitation programme
* Being able to walk before suffering the stroke
* Having the ability to understand and follow simple instructions
* Being hemodynamically stable within the first week after stroke

Exclusion Criteria:

* Poor vital prognosis
* Pathologies or disorders hampering the development of the study such as: blindness, prosthetics, sensory disorders, severe cognitive impairment and so on
* Absence of motor impairments after stroke
* Pre-stroke disorders that affected the ability to walk

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Barthel Index | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Viosca-Herrero, PhD, Study Director — Hospital Universitario La Fe; Juan-Manuel Belda-Lois, PhD, Study Director — Instituto de Biomecanica de Valencia; Celedonia Igual-Camacho, PhD, Study Director — University of Valencia
Locations (1):
- Hospital La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Sanchez-Sanchez ML, Belda-Lois JM, Mena-Del Horno S, Viosca-Herrero E, Igual-Camacho C, Gisbert-Morant B. A new methodology based on functional principal component analysis to study postural stability post-stroke. Clin Biomech (Bristol). 2018 Jul;56:18-26. doi: 10.1016/j.clinbiomech.2018.05.003. Epub 2018 May 5. PMID 29775954